CLINICAL TRIAL: NCT02108977
Title: Evaluation of Videoconferencing vs Telephone Genetic Counseling Consultations
Brief Title: Evaluation of Videoconferencing Versus Telephone Genetic Counseling
Acronym: EVTGC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: PPO 13-364
Record Dates: First submitted 2014-03-31; First posted 2014-04-09 (Estimated); Results first posted 2016-04-21 (Estimated); Last update posted 2019-03-28 (Actual); Status verified 2019-03

CONDITIONS: Remote Consultation, Teleconsultation; Remote Consultation, Video
Keywords: Remote Consultation; Teleconsultation; Videoconferencing; Genetic Counseling; Costs and Cost Analysis; Comparative Effectiveness Research; Telehealth

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Videoconferencing Genetic Consultation (Experimental): Patients will travel to CBOC and receive genetic counseling session via videoconferencing
  Interventions: Other: Videoconferencing Genetic Consultation
- Teleconferencing Genetic Consultation (Active Comparator): Patients will receive genetic counseling session via telephone (usual treatment)
  Interventions: Other: Teleconferencing Genetic Consultation

INTERVENTIONS:
Other: Videoconferencing Genetic Consultation — Patients will travel to CBOC and receive genetic counseling session via videoconferencing
  Arms: Videoconferencing Genetic Consultation
Other: Teleconferencing Genetic Consultation — Patients will receive genetic counseling session via telephone (usual treatment)
  Arms: Teleconferencing Genetic Consultation

SUMMARY:
Genetic counseling has benefits for individuals and their family members in their health care decision-making. Provision of genetic counseling has been deemed standard of care by several medical organizations and incorporated into clinical guidelines, such as those of the US Preventive Services Task Force. To better comply with these guidelines, Genomic Medicine Service (GMS) recently established at the Salt Lake City, Utah VA medical center to provide genomic services and counseling as a part of VA Patient Care Services. For Veterans for whom in-person genetic counseling in not feasible, GMS conducts counseling either via telephone or videoconferencing. Although both of these methods can be effective for delivering genetic counseling, each has its relative advantages and disadvantages. The specific aim of this study is to gain a better understanding of the advantages and disadvantages of these two modalities. This information will be useful not only for genetic counseling but also other interventions that use telephone or videoconferencing to access patients.

DETAILED DESCRIPTION:
Objectives: This is a Type 1 hybrid pre-implementation study whose specific aims are to: 1) Compare retention of genetic counseling information provided to patients via telephone versus videoconferencing; 2) Use validated surveys to quantitatively assess satisfaction with genetic counseling conducted via telephone versus videoconferencing; 3) Conduct interviews with patients to qualitatively assess positive and negative aspects of their experience, barriers, and facilitators with genetic counseling via telephone or videoconferencing; 4) Conduct interviews with the genetic counselors at Genomic Medicine Service (GMS) to qualitatively assess barriers and facilitators to conducting genetic counseling via telephone and videoconferencing; and 5) Conduct a cost analysis of the telephone and videoconferencing genetic counseling modalities.

Methods: We will undertake a randomized controlled trial of Veterans that are willing to have genetic counseling conducted either via telephone or videoconferencing. Veterans with multiple polyps referred to GMS for genetic counseling will undergo a screening interview by telephone to obtain information about personal and family history and study inclusion and exclusion criteria eligibility. If criteria are met, they will be given information about the study and asked to provide informed consent. If consent is provided, baseline questions will be asked to collect demographic information and assess genetic knowledge. Randomization via random number generation will be used to assign subjects to either the telephone or videoconferencing arms. Lastly, a genetic counseling session will be scheduled for each patient.

Within one week of receiving genetic counseling, participants will be called to assess knowledge retention, conduct the satisfaction surveys and numeracy, and to schedule the qualitative interview for the subset of patients (10-12 per study arm) who agree to participate. We will use the Consolidated Framework for Implementation Research to develop and conduct qualitative interviews with the GMS staff.

Based on power calculation, we will need a sample size of 56 subjects. To achieve this sample size we will need to recruit approximately two to three subjects per week over a seven month period. This requires a reasonable participation rate between 32-40% of polyposis patients referred to GMS for genetic counseling.

Data analysis will begin with descriptive statistics to describe our study sample. To assess differences in knowledge retention and satisfaction between the telephone and videoconferencing groups, we will use Chi-square test for categorical variables and the Wilcoxon-rank sum test for discrete ordinal and continuous variables. We will also conduct multivariable ordinary least squares regression to assess whether knowledge retention or satisfaction differs according to patient characteristics, numeracy, or genetic counselor. The qualitative interviews will be digital audio recorded and transcribed for analysis. We will use a directed approach to content analysis. Analysis will be conducted with Atlas.ti qualitative analysis software that facilitates management of coding and analysis of patterns across transcripts. Cost analysis of the two counseling options will be assessed by direct measurement of equipment and labor input costs as well as travel reimbursement by the VA. From the patient's perspective, the costs associated with traveling to a VA clinic site with videoconferencing equipment will also be considered.

ELIGIBILITY:
Inclusion Criteria:

* Age 50 or greater,
* a finding of 10 or more lifetime adenomatous polyps or sessile polyps,
* no contributing family history,
* and the patient must be able to be reached by telephone and speak English

Exclusion Criteria:

* Complex family history (family members with other cancers) or one suggestive of a known colon cancer syndrome,
* unwillingness to travel to a VA site with videoconferencing capability,
* diagnosis of colon cancer

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2014-04; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Santanu K. Datta, PhD, Principal Investigator — Durham VA Medical Center, Durham, NC
Locations (2):
- United States (2):
  - Durham VA Medical Center, Durham, NC, Durham, North Carolina
  - VA Salt Lake City Health Care System, Salt Lake City, UT, Salt Lake City, Utah

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Videoconferencing Genetic Consultation | Teleconferencing Genetic Consultation
Started | 18 | 20
Completed | 8 | 19
Not Completed | 10 | 1

BASELINE CHARACTERISTICS:
Population: We define baseline participants as those who enrolled in the study and participated in the knowledge pre-test.
Groups:
- Telephone Genetic Consultation: Patients will receive genetic counseling session via telephone (usual treatment)
  Teleconferencing Genetic Consultation: Patients will receive genetic counseling session via telephone (usual treatment)
- Total: Total of all reporting groups
Arm/Group | Videoconferencing Genetic Consultation | Telephone Genetic Consultation | Total
Number analyzed (Participants) | 8 | 19 | 27
Age, Customized [Number; unit: Not collected] — Age data was not collected
  Not collected | NA — Age data was not collected | NA — Age data was not collected | NA — Total not calculated because data are not available (NA) in one or more arms.
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 8 | 19 | 27

OUTCOME MEASURES:

1. Primary Outcome: Assessment of Knowledge Retention of Genetic Counseling Information Via 8-Question Pre- and Post-Counseling Assessment
Description: Subjects will be asked 8 True/False genetics-related questions before and after counseling to assess improvement and retention of genetic counseling knowledge and information
Time Frame: Pre- and post- (within 2 weeks) genetic counseling
Measure: Mean (Standard Deviation); unit: Number of correct answers (out of 8)
Arm/Group | Videoconferencing Genetic Consultation | Teleconferencing Genetic Consultation
Number analyzed (Participants) | 8 | 19
Number of correct answers (out of 8)
  Correct Answers Pre-Consultation | 5.63 (1.19) | 4.37 (1.54)
  Correct Answers Post-Consultation | 6.50 (0.93) | 4.74 (1.19)

2. Primary Outcome: Satisfaction With Genetic Counseling Session Using the Genetic Counseling Satisfaction Scale
Description: 6-question Genetic Counseling Satisfaction Scale using 5-point Likert scale responses Strongly Disagree (1) to Strongly Agree (5)
Time Frame: Within two weeks of receiving genetic counseling
Measure: Mean (Standard Deviation); unit: points on a scale of 30 (most satisfied)
Arm/Group | Videoconferencing Genetic Consultation | Teleconferencing Genetic Consultation
Number analyzed (Participants) | 8 | 19
points on a scale of 30 (most satisfied) | 26.88 (3.04) | 25.21 (2.64)

3. Primary Outcome: Qualitative Assessment of Genetic Counseling Experience, Barriers and Facilitators by PATIENTS
Description: We asked the subjects to discuss specific aspects of each modality including the ease of use, navigation, and adaptability of each modality, conveying and comprehending genetic and numeric information, and perceived advantages and disadvantages of each modality.
Time Frame: Within six weeks of receiving genetic counseling
Population: A subsample of patients in each modality was interviewed to qualitatively assess the satisfaction with the counseling they received, and the benefits and limitations of the modality, whether it was by phone or video.
Measure: Number; unit: participants
Arm/Group | Videoconferencing Genetic Consultation | Teleconferencing Genetic Consultation
Number analyzed (Participants) | 7 | 6
participants | NA — The data is qualitative in nature collected via interview | NA — The data is qualitative in nature collected via interview

4. Primary Outcome: Qualitative Assessment of Genetic Counseling Experience, Barriers and Facilitators by GENETIC COUNSELORS
Description: Five counselors agreed to be interviewed. We asked them to discuss specific aspects of each modality including the ease of use, navigation, and adaptability of each modality, conveying and comprehending genetic and numeric information, and perceived advantages and disadvantages of each modality.
Time Frame: Within 4 weeks after study data collection was completed
Population: A subsample of counselors in each modality was interviewed to qualitatively assess the satisfaction with the counseling they provided, and the benefits and limitations of the modality, whether it was by phone or video.
Measure: Count of Participants; unit: Participants
Groups:
- Videoconferencing Genetic Consultation: Counselors provided genetic counseling via videoconferencing.
- Teleconferencing Genetic Consultation: Counselors provided genetic counseling via telephone.
Arm/Group | Videoconferencing Genetic Consultation | Teleconferencing Genetic Consultation
Number analyzed (Participants) | 5 | 5
Participants | NA — Data is qualitative in nature and collected via interview. | NA — Data is qualitative in nature and collected via interview.

5. Primary Outcome: Cost Analysis
Description: Labor (including training) and non-labor (e.g., equipment cost) inputs required to provide counseling via telephone versus videoconferencing. Patient travels costs will be included via self-report.
Time Frame: Cost analysis will be conducted in months 10-12 of grant period (projected January 1-March 31, 2015)
Population: Travel distance data not applicable to the Teleconferencing group.
Measure: Median (Inter-Quartile Range); unit: Loss of Productivity Cost in US Dollars
Arm/Group | Videoconferencing Genetic Consultation | Teleconferencing Genetic Consultation
Number analyzed (Participants) | 8 | 0
Loss of Productivity Cost in US Dollars | 67.29 [44.78 to 97.88] |

ADVERSE EVENTS:
Description: There were no participants affected by any serious Adverse Events
Arm/Group | Videoconferencing Genetic Consultation | Teleconferencing Genetic Consultation
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/19
Other Adverse Events (participants affected / at risk) | 0/8 | 0/19

LIMITATIONS AND CAVEATS:
We did not achieve the study sample that we hoped to achieve. Patients randomized to the telephone arm participated in the study, whereas patients randomized to the videoconferencing arm often dropped out of the study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes